CLINICAL TRIAL: NCT06030596
Title: SPECT Myocardial Blood Flow Quantification for Diagnosis of Ischemic Heart Disease Determined by Fraction Flow Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Wei Fang, MD, China National Center for Cardiovascular Diseases
Other Study IDs: SPECT MBFQ Trial II
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
Keywords: SPECT; Myocardial Blood Flow; Myocardial Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- coronary artery disease: Suspected or known coronary artery disease

SUMMARY:
Recent evidences have demonstrated improved diagnostic accuracy for detecting coronary artery disease (CAD) when myocardial blood flow (MBF) is quantified in absolute terms using single photon emission tomography (SPECT) compared to conventional myocardial perfusion imaging (MPI). However, there are no uniformly accepted cutoff values of MBF and MFR derived from SPECT for diagnosing hemodynamically significant CAD. Particularly, the diagnostic performance for quantitative SPECT has not been validated using fractional flow reserve (FFR). The aim of this prospective study is to determine optimal cutoff values of absolute MBF and MFR derived from NaI (Tl)-based SPECT and to evaluate the diagnostic efficacy of this quantitative technology utilizing invasive coronary angiography (ICA) in combination with FFR results as the reference standard in patients with suspected or known CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 79 years old
* At least one CAD risk factor
* Intermediate to high pre-test likelihood for CAD
* Suspected or known CAD, clinically referred for invasive coronary angiography
* Able and willing to comply with the study procedures
* Written informed consent

Exclusion Criteria:

* History or risk of severe bradycardia
* History of myocardial infarction, dilated cardiomyopathy, hypertrophic cardiomyopathy, valve issue or congenital heart disease
* Wheezing asthma or COPD
* Known second- or third-degree AV block
* Known hypersensitivity to dipyridamole or adenosine
* Known coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) prior to screening
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or known CAD
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of MBF and MFR derived from SPECT | 1 year
  The diagnostic sensitivity, specificity, accuracy of MBF and MFR derived from SPECT for the detection of hemodynamically significant coronary artery disease as defined by invasive coronary angiography in combination with fractional flow reserve measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD/PhD, Study Chair — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No